CLINICAL TRIAL: NCT01519115
Title: A Comparison of Clinic Outcomes Between Early Physical Therapy Intervention and Usual Care in Individuals Following Anterior Cervical Fusion
Brief Title: Comparison of Outcomes Between Early Physical Therapy Intervention and Usual Care Following Anterior Cervical Fusion Surgery
Acronym: ACF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Society of Allied Health Professions (Unknown); Texas Spine and Joint Hospital (Unknown)
Responsible Party: Principal Investigator, cmcfarland, Carol McFarland PT, MS, doctoral student, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16841
Record Dates: First submitted 2012-01-19; First posted 2012-01-26 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Cervical Spine Degenerative Disc Disease; Fusion of Spine, Cervical Region
Keywords: deep cervical flexors; spine stabilization; posture; function; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): usual care of one physical therapy visit in hospital after ACF surgery
  Interventions: Other: usual care
- Early physical therapy intervention (Experimental): early physical therapy program instructed and followed at home for 6 weeks
  Interventions: Other: early physical therapy intervention

INTERVENTIONS:
Other: early physical therapy intervention — instruction in home care program to be followed for first six weeks after ACF surgery
  Other Names: cervical spine stabilization; posture training; perioperative spine care
  Arms: Early physical therapy intervention
Other: usual care — one physical therapy visit in hospital following ACF surgery
  Other Names: post operative spine precautions; perioperative spine care
  Arms: Usual care

SUMMARY:
Background: Early physical therapy (PT) intervention with emphasis on spinal stabilization has been shown to benefit individuals undergoing lumbar spinal surgery. Further, training cervical spine stabilizers (deep cervical flexors and cervical multifidus) has been shown to be effective in reducing neck pain, restoring cervical spinal function and mobility in many types of cervical spine dysfunction. However, the training of stabilizers has not been studied in individuals undergoing cervical spinal surgery, even though these individuals often have problems with residual pain and weakness after the surgery.

Purpose: The purpose of this study is to compare the effectiveness of clinical outcomes between an early PT intervention and usual care in patients who have undergone anterior cervical spine fusion (ACF) surgery. A study hypothesis is that outcomes will be improved with early PT intervention.

Methods: This study is a double-blinded randomized clinical trial with a two-factor (2x3) research design. The patients following ACF surgery will be randomly assigned in one of the two treatment groups: usual care and early intervention. Three outcome measures will be collected pre-operative for baseline, and then at 6-week and 12-week post-operative follow-up visits, including: (1) deep cervical flexor (DCF) strength as determined by the cranio-cervical flexion (CCF) performance test, (2) patient's perceived disability associated neck pain as determined by the Neck Disability Index (NDI) questionnaire, and (3) neck pain level using the numeric pain rating scale (NPRS). In addition, at 6 and 12 weeks, the global rate of change (GROC) scale will be obtained to determine the patient's perception of overall improvement as a result of surgery. The investigator performing the outcome measures will be blinded to group assignment, and therefore will not participate in treatment. After randomization, the usual care group will receive only one visit of PT for post-operative instruction. The early intervention group will receive verbal and written instructions for posture and training cervical spine stabilizers in addition to the usual care. The early intervention group also will be asked to perform these exercises at home and keep a log of the exercise.

Data Analysis: Two 2x3 MANOVAs with repeated measures will be used to examine the differences in the CCF strength and the NDI scores between groups and at the three different time frames with the α level set at 0.05. Non-parametric tests (Mann-Whitney U tests) will be used to compare the differences in the NPRS and GROC data over time and between groups.

DETAILED DESCRIPTION:
Study Enrollment A research assistant will enroll participants, obtain informed consent, and randomly assign participants to the two groups. Therefore, the research assistant will not be blinded to group assignment. The primary investigator (PI) will perform all clinical tests, and will be blinded to group assignment, and therefore will not perform the PT interventions. Three licensed PTs will be trained in both usual care and early PT interventions. The research assistant will inform the PT assigned to each study participant of group assignment and provide materials for treatment.

Clinical Examination All participants will undergo a neurological examination for cervical spine, including light touch sensory testing, muscle testing, deep tendon reflex testing, and neural tension testing of upper extremities in order to identify neurologic deficits. These clinical tests will be performed pre-operatively and at 6 and 12 weeks post-operatively. During post-operative visits, operative reports and post-operative radiographs will also be collected to identify complications from the surgery that may affect the study results, but will not be used in determining outcome measures.

Clinical Outcome Measurements and Instruments

1. Cranio-cervical Flexor Strength (CCF-S) Testing The CCF-S test will be used to determine DCF strength using the StabilizerTM Pressure Biofeedback (Chattanooga Group, Inc, Chattanooga, TN) (see Appendix A). The investigator will ask the participants to lie in a supine position with knees flexed and the Stabilizer placed under the neck so that it supports the cervical spine from just below the occiput to the cervical-thoracic junction. The cuff will then be inflated to 20 mm Hg. to support the cervical spine without adding anterior forces to the vertebrae. The investigator will instruct the participant to do a slight nodding movement, a chin-tuck, producing enough additional pressure on the cuff to increase the pressure to 22 mmHg. The participant will be asked to hold the pressure at this level for 10 seconds. If they are able to perform this successfully, the participant is then asked to try to increase the pressure to 24 mm Hg for 10 sec., and if successful, increase to 26 mm. They will proceed in 2 mm increments up to a maximum of 30 mmHg. The highest pressure that the participant is able to hold for 10 seconds is defined the CCF-S score. The participants will perform the CCF-S test twice and the better of two trials will be used for data analysis. The reliability and validity of the test has been established on individuals with and without neck pain symptoms.
2. Cranio-cervical Flexor Endurance (CCF-E) Testing The endurance test for the DCF is performed by asking the participant to hold the pressure of the CCF-S test for 10 seconds up to a maximum of 10 repetitions. This test will be stopped on the repetition where the participant fails to hold the target pressure on the Stabilizer. Only the successful repetitions will be counted, and that number multiplied by ten will be the CCF-E score. If the participant is observed to use substitute motions or activate superficial neck flexors, they will also be stopped. The CCF-E will be determined with a single trial in this study.
3. Neck Pain Disability Index (Appendix C) The Neck Pain Disability Index (NDI) will be used to determine the patient's perceived disability associated with neck pain. The NDI is a commonly used scale with 10 items assessing level of neck function. The NDI has been shown to be reliable and valid in several studies.
4. Numeric Pain Rating Scale The Numeric Pain Rating Scale (NPRS) will be used to determine the patient's pain level. The NPRS is a well known scale from 0-10 used in many medical settings for patients to rate their level of pain.
5. Global Rating of Change scale The Global Rating of Change (GROC) scale will be used to determine the patient's perception of overall improvement. The GROC is a 15-point numerical scale from -7 (much worse) through 0 (no change) to +7 (much better), for patients to rate the amount of change since surgery. This scale will only be given to participants at the two post-operative time frames.

Intervention The three PTs who will administer physical therapy for the in-patient stay following ACF, will be trained to standardize the treatment protocols of both the usual care and early PT intervention. After the participant is randomly assigned to one of the two groups, the PTs will receive a packet with the materials needed for the assigned group for this participant from the research assistant.

1. Usual Care Group For participants in the usual care group, the intervention will closely follow current common practice in the first 6 weeks post-operatively for patients after ACF. These participants will be seen in the hospital by one of the two treating PTs before discharge. The participants will be instructed the Patient Information Sheet on ACF. They will also view the DVD titled "First Six Weeks", a summary of the general post spine surgery precautions. The treating PT will address any questions on the video, and evaluate the participant for proper positioning of head and neck, use and fit of cervical collar if applicable, proper body mechanics, and safety with transfers and gait. In the patient instructions for ACF, patients are encouraged to pay attention to good posture, and work on walking increasing distances to help the fusion. However, they are not given any means of recording or tracking their progress with walking distance.
2. Early Physical Therapy Intervention Group The participants in the early PT intervention group will receive the same instruction as the usual care group. In addition, they will be instructed in a series of exercises referred to as "Postural and Neck Protection Training" with attention to head positioning and recruiting cervical segmental stabilizers, i.e. DCF, and postural muscles. They will be instructed in controlling pain that may occur with the exercises. Strategies for pain control will include head and shoulder posture correction, position and support of the entire spine such as lumbar support, ice application, deep breathing and relaxation techniques. The participants will be given specific instructions on exercise and activity with a home exercise log in which they can record daily practice of the exercise program and the time spent walking.

Follow-up calls to all participants will be conducted by a research assistant at 2 and 4 weeks post surgery to verify compliance with the program and address any questions. Questions that require help from the PT will be relayed to the principle investigator (PI) without identifying the participant.

All participants in both groups will also be encouraged to call the assistant with any questions throughout the study. Questions will be relayed from the assistant to the PI, so that the PI will remain blinded to group assignment.

Reliability Testing Although the CCF tests have had reliability established for individuals with and without neck pain, reliability has not been established for individuals who have undergone cervical spine surgery. Therefore, same-day reliability will be tested on the first ten participants who are able to complete the CCF-S and CCF-E test at the 6-week post-operative data collection. These individuals will perform the CCF-S tests twice, at the beginning and the end of their testing session to allow rest in between. Therefore, the CCF will be the first outcome measure completed, followed by the other clinical measures. For between-day reliability, participants who live in close proximity to the hospital will be measured again with a brief return visit for a second time for repeating the CCF tests.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the age of 30 to 70 years
2. Individuals who have consulted one of the five participating spine surgeons and are scheduled for ACF surgery at Texas Spine and Joint Hospital
3. Surgical candidates classified as Task Force category III, with neurologic deficit without major structural pathology, or IV, with major structural pathology -

Exclusion Criteria:

1. Musculoskeletal or systemic disorders with functional impairments that will limit tolerance of testing.
2. Pain greater than 8/10 on the NPRS that often indicates severe pathology and therefore limits testing tolerance.
3. Prior cervical spine surgeries.
4. More than two level cervical spine surgery planned. -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in cranio-cervical flexor strength from before surgery to 6 and 12 weeks post operative | during preo-perative medical exam 1-2 weeks before surgery, and 6 and 12 weeks post
  test described in protocol information

SECONDARY OUTCOMES:
Change in Neck Disability Index from pre-operative condition to 6 and 12 weeks post operative | during pre-operative medical exam 1-2 weeks before surgery and 6 and 12 weeks post
  test described in protocol description

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang, PT, PhD, Study Chair — Texas Woman's University; Carol McFarland, PT, MS, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Spine and Joint Hospital, Tyler, Texas, United States

REFERENCES:
- [Background] Abbott AD, Tyni-Lenne R, Hedlund R. Early rehabilitation targeting cognition, behavior, and motor function after lumbar fusion: a randomized controlled trial. Spine (Phila Pa 1976). 2010 Apr 15;35(8):848-57. doi: 10.1097/BRS.0b013e3181d1049f. PMID 20354468
- [Background] Peolsson A, Kjellman G. Neck muscle endurance in nonspecific patients with neck pain and in patients after anterior cervical decompression and fusion. J Manipulative Physiol Ther. 2007 Jun;30(5):343-50. doi: 10.1016/j.jmpt.2007.04.008. PMID 17574951
- [Background] Ylinen JJ, Savolainen S, Airaksinen O, Kautiainen H, Salo P, Hakkinen A. Decreased strength and mobility in patients after anterior cervical diskectomy compared with healthy subjects. Arch Phys Med Rehabil. 2003 Jul;84(7):1043-7. doi: 10.1016/s0003-9993(03)00039-x. PMID 12881832
- [Background] O'Leary S, Falla D, Elliott JM, Jull G. Muscle dysfunction in cervical spine pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):324-33. doi: 10.2519/jospt.2009.2872. PMID 19411767
- [Background] Chiu TT, Law EY, Chiu TH. Performance of the craniocervical flexion test in subjects with and without chronic neck pain. J Orthop Sports Phys Ther. 2005 Sep;35(9):567-71. doi: 10.2519/jospt.2005.35.9.567. PMID 16268243
- [Background] Johansson AC, Linton SJ, Bergkvist L, Nilsson O, Cornefjord M. Clinic-based training in comparison to home-based training after first-time lumbar disc surgery: a randomised controlled trial. Eur Spine J. 2009 Mar;18(3):398-409. doi: 10.1007/s00586-008-0826-3. Epub 2008 Nov 20. PMID 19020904
- [Derived] McFarland C, Wang-Price S, Gordon CR, Danielson GO, Crutchfield JS, Medley A, Roddey T. A Comparison of Clinical Outcomes between Early Cervical Spine Stabilizer Training and Usual Care in Individuals following Anterior Cervical Discectomy and Fusion. Rehabil Res Pract. 2020 Apr 24;2020:5946152. doi: 10.1155/2020/5946152. eCollection 2020. PMID 32373366